CLINICAL TRIAL: NCT04282759
Title: Difficulty in Laparoscopic Cholecystectomy Score Can Determine the Operative Challenge.
Brief Title: Can Laparoscopic Cholecystectomy Difficulty Score Predict Difficult Surgery
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Erguvan Nalıncıoğlu, principal investigator, Konya Meram State Hospital
Other Study IDs: KonyaHPRC
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Laparoscopic cholecystectomy is the gold standard treatment method in symptomatic gallstone disease. However, complications that develop due to being a technical procedure tend to be more complex and more morbid-estimating how difficult the surgery will be before the operation will enable us to be more prepared both in terms of patient counseling and surgical team selection. Such a prediction will minimize the risk of complications and morbidity.

In our study, investigators used the scoring system "How to predict difficult laparoscopic cholecystectomy? Proposal for a simple preoperative scoring system?" which was published in "The American Journal of Surgery" in November 2016. Investigators wanted to evaluate prospectively adequate "Laparoscopic Cholecystectomy Difficulty Score," which was developed retrospectively, in determining the surgical difficulty preoperatively.

DETAILED DESCRIPTION:
ETHICAL BOARD APPROVAL

Konya Chamber of Commerce Education and Health Foundation was found ethically appropriate for the study according to the decision of Karatay University Ethical Board Presidency dated 18.06.2019 and numbered 2019/0051.

FEATURES OF THE STUDY AND SELECTION OF PATIENTS

Patients who were to be operated due to symptomatic cholelithiasis between 01.03.2020 and 31.07.2020 at the Health Sciences University (SBU) Konya Training and Research Hospital (KEAH) were included in the study. The study was done prospectively.

Laparoscopic Cholecystectomy Difficulty Score (DSLC) developed in the reference study will be used. The sex of the patients and whether they had an attack of cholecystitis will be recorded. Neutrophil count, fibrinogen, and ALP levels will be recorded from preoperatively routine blood tests. DSLC score will be calculated before the patient goes into surgery. How successful the scoring system is in determining the difficulty of the operation in the postoperative period will be analyzed statistically.

Thirteen surgeons will be included in the study. Based on the last ten surgery times, where each surgeon has no problems and has no technical difficulties, the average operation time will be calculated for each surgeon individually. In the reference study, it has been accepted that the surgeon's duration is more than 1.5 times or challenging to undergo open surgery. In our study, it will be considered as a difficult operation to exceed or exceed 1.5 times the surgeon's duration. Other than that, it will be considered a smooth operation. The biliary tract injuries that occurred in exposed cases will be classified according to the Strasberg classification. In the reference study, statistically significant score groups were formed as low risk of 0 points, medium risk of 1-4 points, high risk of 5-9 points, and a very high risk of 10 points. In our study, these score groups will be created, and statistical analysis will be made. Also, ROC (Reciever Operator Characteristics Curve) curve will be created with the scores obtained from the scoring system, and the specificity and sensitivity of the scoring system will be statistically put.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be operated for biliary colic, chronic cholecystitis or symptomatic cholelithiasis,
* Patients who have been treated with antibiotics before with the diagnosis of cholecystitis and have been planned for elective cholecystectomy,
* Patients diagnosed with acute cholecystitis according to Tokyo criteria and cholecystectomy planned due to acute cholecystitis

Exclusion Criteria:

* Patients under the age of 18,
* Patients over 100 years old,
* Patients diagnosed with choledocholithiasis with magnetic resonance cholangiopancreatography (MRCP),
* Patients with cholangitis
* Patients who have undergone endoscopic retrograde cholangiopancreatography (ERCP),
* Patients who have undergone biliary system intervention before,
* Patients scheduled for operation open cholecystectomy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of patients between the ages of 18-100, who are referred to the general surgery clinic for laparoscopic cholecystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Numerical recording of Difficulty Score of Laparoscopic Cholecystectomy (DSLC) | The period of the study is between 1 March 2020 and 15 August 2020.
  Laparoscopic cholecystectomy scores of patients included in the study will be recorded. The relationship between the scoring system and the fact that the cases are easy or difficult will be analyzed statistically, in which predictive values determine the difficulty of the operation. The study will be terminated with the completion of the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bourgouin S, Mancini J, Monchal T, Calvary R, Bordes J, Balandraud P. How to predict difficult laparoscopic cholecystectomy? Proposal for a simple preoperative scoring system. Am J Surg. 2016 Nov;212(5):873-881. doi: 10.1016/j.amjsurg.2016.04.003. Epub 2016 Jun 1. PMID 27329073
- [Background] Sugrue M, Coccolini F, Bucholc M, Johnston A; Contributors from WSES. Intra-operative gallbladder scoring predicts conversion of laparoscopic to open cholecystectomy: a WSES prospective collaborative study. World J Emerg Surg. 2019 Mar 14;14:12. doi: 10.1186/s13017-019-0230-9. eCollection 2019. PMID 30911325